CLINICAL TRIAL: NCT04614272
Title: The Effect of Praying on Endogenous Pain Modulation and Pain Intensity in Healthy Religious Individuals: A Randomized Controlled Experiment
Brief Title: Effect of Prayer on Conditioned Pain Modulation and on Pain Intensity in Healthy Religious University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonine University (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, charbel najem, assisstant professor, Antonine University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: charbel najem
Record Dates: First submitted 2020-10-20; First posted 2020-11-03 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Faith Healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: while assessing for endogenous pain inhibition and pain intensity the assessor will be blind and will not know to which group the participant belong. Participants will be blinded by being blind to the study hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active prayer group (Experimental): the active prayer group will mediate over an active type of prayer
  Interventions: Behavioral: Prayer
- passive prayer group (Experimental): the passive prayer group will mediate over a passive type of prayer
  Interventions: Behavioral: Prayer
- control group (Sham Comparator): the control group will read a poem
  Interventions: Behavioral: Reading a poem

INTERVENTIONS:
Behavioral: Prayer — Prayer is a non-pharmaceutical method of pain management and a form of alternative medicine.
  Arms: active prayer group; passive prayer group
Behavioral: Reading a poem — Reading is a distraction tool for pain management
  Arms: control group

SUMMARY:
With this study the investigators wish to examine the effect of prayer on pain intensity and on the conditioned pain modulation in healthy religious university students.

DETAILED DESCRIPTION:
There has been a call for a model that incorporate spirituality in the biopsychosocial framework .The biopsychosocial- spiritual model recognizes the impact of the religious factors in modulating the biology of pain.

The aim of this study is to measure the effect of praying as an intervention on conditioned pain modulation and on pain intensity.

The investigators hypothesize that prayer would increase conditioned pain modulation compared to a no prayer control group in a healthy religious population.

The investigators hypothesize that participants engaging in active prayer will show a higher increase in conditioned pain modulation compared to those engaging in passive prayer or no prayer.

The present study is a randomized controlled trial comparing the effect of two types of prayer, the passive and the active prayer and no prayer, on conditioned pain modulation using the heat protocol and on pain intensity. Participants are to be randomly assigned to 2 groups: the prayer group and the control group.

The control group is of (n=50) participants and the prayer group is (n=150) participants to be divided according to the style of praying identified by the prayer function scale into active and passive prayer group.

Appropriate statistical analyses will be performed to evaluate and compare treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female.
* Healthy male.
* University students
* Religious participants who would score at least two over six on the Non Organizational Religious Activities subscale of the Duke University Religious Index.

Exclusion Criteria:

* Pregnant women.
* Individuals with chronic pain.
* Individuals with psychiatric disease.
* Individuals suffering from headache for more than 2 days a month.
* Individuals with high blood pressure.
* Individuals under regular use of medication.
* Individuals who would score 1 or 0 on the on the Non Organizational Religious Activities subscale of the Duke University Religious Index.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
change in conditioned pain modulation (CPM) | Measured prior to intervention (baseline=day 1) and immediate following the intervention (=day 1)
  the conditioned pain modulation paradigm (pressure pain threshold using a digital algometer as test stimulus and the heat pressor test (immersion of one hand in hot water of 45.5°C) as conditioning stimulus
change in pain intensity | Measured prior to intervention (baseline=day 1) and immediate following the intervention (=day 1)
  numeric rating scale from 0 to 100 where 0 is no pain and 100 is the worst pain imaginable

SECONDARY OUTCOMES:
The Duke University Religion Index | religiosity is assessed at baseline
  1.The religiosity level will be measured using the Duke University Religiosity scale, it is a 5-item self-report measure of religious involvement scored on a 5-point Likert-type scale ranging from 1 (almost never) to 5 (a great deal). It assesses the three major dimensions of religiosity, organizational religious activity, non-organizational religious activity, and intrinsic religiosity .
Prayer function scale | the prayer function scale is assessed at baseline
  is a self-report instrument that assesses the motivation or purpose behind an individual's prayer while she or he is coping with difficult circumstances.
  The scale consists of 58 items that are scored on a 5-point Likert-type scale ranging from 1 (almost never) to 5 (a great deal).
  The measure contains four scales: Provides Acceptance (17 items), Provides Calm and Focus (11 items), Deferring/Avoiding , and Provides Assistance (14 items).
  The deferring/avoiding scale represent a passive type of prayer The assistance scale represent an active type of prayer.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Meeus, Phd, Study Director — University Ghent
Locations (1):
- Antonine University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
the data will only be used for this study